CLINICAL TRIAL: NCT00775801
Title: An IDE Study of the Freedom Lumbar Disc in the Treatment of Lumbar Degenerative Disc Disease
Brief Title: Freedom Lumbar Disc in the Treatment of Lumbar Degenerative Disc Disease
Acronym: FLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AxioMed Spine Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-125
Record Dates: First submitted 2008-10-13; First posted 2008-10-20 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Degenerative Disc Disease (DDD)
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): FLD
  Interventions: Device: FLD
- Control (Active Comparator)
  Interventions: Device: Control

INTERVENTIONS:
Device: FLD — Artificial lumbar disc
  Arms: Treatment
Device: Control — Artificial lumbar disc
  Arms: Control

SUMMARY:
This study will look at the result of using the FLD device as an artificial lumbar disc. The study will compare the safety and effectiveness of the FLD artificial lumbar disc to an already approved artificial lumbar disc.

DETAILED DESCRIPTION:
The Freedom Lumbar Disc is indicated for spinal arthroplasty in skeletally mature patients with single level, symptomatic degenerative disc disease (DDD) from L3-S1. This is a prospective, multi-center, randomized, controlled trial. Subjects with DDD will be randomized to disc arthroplasty with the FLD device or a control device. The overall purpose (objective) of this trial is to collect clinical data to demonstrate the safety and effectiveness of FLD used for the treatment of symptomatic lumbar degenerative disc disease compared to the control device.

ELIGIBILITY:
Inclusion Criteria:

* Single level, degenerative disc disease at L3 to S1, inclusive.
* Minimum of 6 months of unsuccessful conservative treatment.
* Subject is a surgical candidate for an anterior approach to the lumbar spine (<3 abdominal surgeries).
* Back pain at the operative level only (by discogram, if necessary).
* Leg pain and/or back pain due to disc space settling, with or without radicular symptoms related to foraminal narrowing.
* Subject must understand and sign the written Informed Consent.

Exclusion Criteria:

* Prior fusion at any lumbar level.
* Clinical evidence of adjacent lumbar segment disease.
* Previous trauma to the L3, L4, L5, or S1 levels (in compression or burst).
* Non-contained or extruded herniated nucleus pulposus.
* Congenital stenosis or central/lateral stenosis (mid-sagittal stenosis of <8mm by CT or MR) secondary to acquired degenerative disease requiring treatment that destabilizes the spine (requiring fusion), or for subjects in whom increased motion may increase symptoms.
* Retro- or spondylolisthesis of ≥ 2.5 mm which is either fixed or present on flexion/extension films, and slippage of vertebral body where the listhesis is due to disc space settling in the absence of degenerative facets or a pars interarticularis defect.
* Significant kyphosis (>11ْ sagittal plane deformity).
* History of any invasive malignancy (except non-melanoma skin cancer) unless treated with curative intent and there have been no clinical signs or symptoms of malignancy for at least 5 years (in particular, spinal tumors).
* Acute or chronic infection (local or systemic).
* Instability or facet joint arthrosis, clinically significant.
* Arachnoiditis.
* Known or suspected allergy to titanium, polyurethane, cobalt, chromium, molybdenum or silicone.
* Radiographic findings of a fused or total collapsed disc.
* Subject using medications or drugs known to potentially interfere with bone or soft tissue healing (high-dose of steroids, osteoclast inhibitors, etc.).
* Systemic disease affecting the spine, including rheumatoid arthritis, autoimmune disease, AIDS, HIV, or hepatitis.
* Paget's disease, osteomalacia or any other metabolic bone disease (excluding osteoporosis which is addressed separately).
* Psychosocial disorders (e.g. evidence or drug or alcohol abuse).
* Morbid (extreme) obesity (BMI ≥ 40 kg/m2).
* Bone growth stimulator use in spine.
* Investigational drug or device use within 30 days.
* Osteoporosis or osteopenia or metabolic bone disease as confirmed by DEXA scan if poor bone quality is suspected (T-score < -1.0).
* If female of childbearing potential, pregnant or interested in becoming pregnant in the next three years.
* Type 1 diabetes, and uncontrolled (or poorly controlled) Type 2 diabetes.
* Subjects with a history of implant rejection.
* Provocative discography with non-concordant pain at the operative level.
* Incarcerated subjects.
* Myelopathy.
* Significant leg pain of a radicular or neurogenic claudication nature.
* Involved vertebral endplates dimensionally smaller then 39 mm in the mediallateral and/or 32 mm in the anterior-posterior directions.
* Subjects not able to meet follow-up requirements.
* Lumbar scoliosis > 11 degrees.
* Any previous or current litigation related to the spine.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-09; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Overall success will be determined by a composite of measures regarding subject self-assessment of function (disability), low back pain, neurological function and device implantation status. | 24 Months

SECONDARY OUTCOMES:
The improvement of subject self-assessment of function (disability), low back pain, patient satisfaction, neurological function and device implantation status at the 24 month follow-up compared to baseline. | 24 Months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - CORE Orthopaedic Medical Center, San Diego, California
  - The Spine Institute, Loveland, Colorado
  - Resurgens Spine Center, Atlanta, Georgia
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Nebraska Spine Center, LLC, Omaha, Nebraska
  - NYU/Hospital for Joint Diseases, New York, New York
  - Carolina NeuroSurgery & Spine Associates, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, P.A., Durham, North Carolina
  - Central Texas Spine Institute, Austin, Texas
  - Texas Back Institute, Plano, Texas
  - Gordon Spine & Brain Associates, Tyler, Texas
- Germany (2):
  - Westend Hospital, Berlin
  - Klinikum-Goerlitz, Görlitz

REFERENCES:
- See also: AxioMed's Website — http://www.axiomed.com